CLINICAL TRIAL: NCT00366652
Title: A Randomized, Open-Label, Crossover, Drug Interaction Study to Evaluate the Effects of DVS SR And Duloxetine on the Pharmacokinetics of Desipramine in Healthy Subjects
Brief Title: Study Evaluating the Effects of DVS SR and Duloxetine on the Pharmacokinetics of Desipramine in Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3151A1-401
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Depression; Depressive Disorder; Depressive Disorder, Major
Keywords: Healthy
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major | interventions — Desipramine; Duloxetine Hydrochloride

INTERVENTIONS:
Drug: desvenlafaxine SR
Drug: desipramine
Drug: duloxetine

SUMMARY:
The purpose of this study is to evaluate the effects of multiple doses of DVS SR and duloxetine on the pharmacokinetics of a single dose of desipramine in healthy subjects.

ELIGIBILITY:
1. Healthy men and women between 18 to 55 years of age.
2. Healthy as determined by the investigator on the basis of medical history and physical examination, laboratory test results, vital signs and a 12-lead electrocardiogram.
3. History of being a nonsmoker for a least 1 year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-09; Study Completion 2006-09

PRIMARY OUTCOMES:
The primary outcome of the study is to evaluate the effects of multiple doses of DVS SR and duloxetine on the pharmacokinetics of a single dose of desipramine in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Neptune City, New Jersey, United States